CLINICAL TRIAL: NCT04083443
Title: Model Development for Pharmacokinetics / Pharmacodynamics of Antimicrobial Drugs in Blood Stream Infections Part 1: Feasibility Study
Brief Title: Model for PK/PD of Antimicrobials in Blood Stream Infection: Feasibility
Acronym: MOBSI1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Collaborators: University of Witten/Herdecke (Other); University of Leipzig (Other); University Hospital Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. Uwe Fuhr, Director, Department I of Pharmacology, University of Cologne
Other Study IDs: MOBSI1
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2019-09

CONDITIONS: Blood Stream Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with blood stream infections: Patients with a high probability of a blood stream infection and an indication for antimicrobial treatment. There will be an additional blood sampling for these patients, which is the only intervention in the study.
  Interventions: Other: Additional blood sampling

INTERVENTIONS:
Other: Additional blood sampling — Blood samples will be taken to assess antimicrobial drug concentrations and microbial DNA blood counts. Per patient, at least 5 and up to 15 samples for drug concentrations and at least 3 and up to 6 samples for DNA counts are taken for a duration of up to 3 days.

SUMMARY:
The current study is a pilot study to assess the feasibility of a superordinate project. The final objective of this superordinate project is to describe and model the pharmacokinetic behaviour of a small number of standard antimicrobials used in the treatment of frequent blood stream infections, and to link this via pharmacodynamic models to (inhibition of) bacterial or fungal growth as well as to clinical outcomes in patients.

DETAILED DESCRIPTION:
Patients with a high probability of a blood stream infection and an indication for antimicrobial treatment will be included. The study comprises the identification of patients as potential study participants, obtaining informed consent, documentation of available potential covariates from patient file, withdrawal of pre-study blood samples (PK, PD, microbiology) including documentation of exact time of sampling and processing of the samples, first drug administration including exact documentation (as part of patient care; not as a study intervention), withdrawal of subsequent blood samples (PK, PD, microbiology) during the next 3 days including documentation of exact time of sampling and processing of the samples, storage of processed samples for further analysis, and, if possible, documentation of patient outcome after 7 days. The following steps are carried out after completion of the clinical part of the study in the individual patient or, when possible, in all patients together or in a subset: Bioanalytics, DNA Counts, assessing primary and secondary study endpoints, pharmacometric analyses including PK parameter estimation, PD parameter estimation and assessment of covariate effects with regard to DNA count, CRP, IL-6 and procalcitonin.

ELIGIBILITY:
Inclusion Criteria:

* High probability of a blood stream infection; this is based on

  * the presence of SIRS [Bone et al. 1992] defined by more than one of the following clinical manifestations:

    1. a body temperature greater than 38°C or less than 36°C
    2. a heart rate greater than 90 beats per minute
    3. tachypnea, manifested by a respiratory rate greater than 20 breaths per minute, or hyperventilation, as indicated by a PaCO2 of less than 32 mm Hg
    4. an alteration in the white blood cell count, such as a count greater than 12,000/µl, a count less than 4,000/µl, or the presence of more than 10 percent immature neutrophils ("bands").

       and
  * the assessment of the treating physician according to the patient's situation that the SIRS is caused by an infection (e.g., patients after treatment with cytotoxic drugs)
* indication for antimicrobial treatment
* Intended use of one of the following antimicrobial agents:

piperacillin/tazobactam; vancomycin; meropenem; ampicillin/sulbactam; flucloxacillin; ceftriaxone; caspofungin (according to the decision of the project coordinator, use of other antimicrobial agents may also be included if anticipated to be used frequently)

* Age: 18 years or older (no upper limit)
* Willing and capable to provide written consent prior to enrolment after ample information has been provided

Exclusion Criteria:

* expected chances to successfully carry out venipunctures to obtain the blood samples required for the study are inadequately low according to the assessment of the physician
* Anemia CTCAE grade >2 (i.e., Hb <8.0 g/dL / 4.9 mmol/L)
* the clinical status of the patients suggests that the anticipated treatment of the patient or other conditions would make participation on the study inappropriate (e.g., terminally ill patients); the respective assessment is done by the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, patients with suspected blood stream infection will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Fraction of eligible patients | Screening
  Fraction of identified and potentially eligible patients willing and able to provide informed consent
Positive blood microbial DNA count | Samples for DNA counts are taken for a duration of up to 3 days.
  Fraction of study participants having any positive blood microbial DNA count for microbes which does not reflect sample contamination
Fraction of patients with at least three samples with microbial DNA | Samples for DNA counts are taken for a duration of up to 3 days.
  Fraction of study participants with at least three samples with quantifiable microbial DNA along with a proper documentation
Plausible time courses of antimicrobial drug concentrations | Samples for antimicrobial drug concentrations are taken for a duration of up to 3 days.
  Fraction of study participants with plausible time courses of antimicrobial drug concentrations along with a proper documentation

SECONDARY OUTCOMES:
Population pharmacokinetic parameters of drugs studied | Samples for antimicrobial drug concentrations are taken for a duration of up to 3 days.
  Pharmacometric analyses including PK parameter estimation
Population pharmacodynamic parameters of drugs studied | Samples for antimicrobial drug concentrations are taken for a duration of up to 3 days.
  Population pharmacodynamic parameters of drugs studied with regard to bacterial DNA count, procalcitonin, IL-6 and C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Uwe D Fuhr, Prof. Dr., Principal Investigator — Institut I für Pharmakologie, University of Cologne, Germany
Locations (4):
- Germany (4):
  - Klinik für Anaesthesiologie, Klinikum der Ludwig-Maximilians-Universität München, Munich, Bavaria
  - Clinical Infectiology, Klinik I für Innere Medizin, University Hospital Cologne, Cologne, North Rhine-Westphalia
  - Klinik für Anästhesiologie und Operative Intensivmedizin Krankenhaus Köln-Merheim Klinikum der Universität Witten/ Herdecke, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Leipzig AöR, Klinik für Gastroenterologie und Rheumatologie, Sektion Hepatologie, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: No